CLINICAL TRIAL: NCT01107340
Title: AMIStem Primary Hip System Prospective Post-marketing Multi-centre Surveillance Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01.004.11
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis; Arthritis; Avascular Necrosis; Fracture of the Femoral Neck or Head; Congenital Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis; Arthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMIStem Hip System (Other): Patients who comply with the protocol and received an AMIStem femoral component.
  Interventions: Device: AMIStem Hip System

INTERVENTIONS:
Device: AMIStem Hip System

SUMMARY:
This is a multicentre post-marketing prospective study to evaluate performance and clinical outcomes of AMIIStem primary hip system.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a good candidate for a primary hip arthroplasty using AMIStem Hip System
* Patient is willing and able to give informed consent to participate in the follow-up program
* Patient is suitable for surgery and able to participate in the follow-up program.
* Those presenting with disease that meets the indication for use for Medacta implants defined in the study (on-label use)

Exclusion Criteria:

* Acute systemic or chronic infection
* Skeletal immaturity
* Severe muscular, neurological, vascular deficiency or other pathologies of the affected limb that may compromise the stability of the implant.
* Bone condition that may compromise the stability of the implant.
* Patient who are unwilling or unable to give consent, or to comply with the protocol and the follow-up program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of implant survivorship using Kaplan Meier curve | 10 years after surgery

SECONDARY OUTCOMES:
Assessment of the patient's physical level of activity using the Oxford Hip Score | pre-op, annually post-op up to 10 years
Assessment of the improvement in quality of life and joint movement using the EuroQol-5D score | pre-op, annually post-op up to 10 years
Assessment of implant survivorship as a measure of safety using Kaplan Meier curve | 6 months, 3 years, 5 years, 7.5 years, 10 years after surgery
Assessment of the clinical outcome following total hip replacement using the Harris Hip Score | pre-op, 6 months, 3 years, 5 years, 7.5 years, 10 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Field, PhD FRCS, Principal Investigator — British Orthopaedic Association
Locations (2):
- Uniklinik Balgrist, Zurich, Switzerland
- The Elective Orthopaedic Centre (EOC), Epsom, Surrey, United Kingdom